CLINICAL TRIAL: NCT04417361
Title: A Pilot Trial of Galcanezumab for Vestibular Migraine
Brief Title: Galcanezumab for Vestibular Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-29340; P0541760 (Other Grant/Funding Number: Eli Lilly and Company)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Vestibular Migraine
Keywords: vestibular migraine; galcanezumab; clinical trial
MeSH Terms: interventions — erenumab

STUDY DESIGN:
Intervention Model Description: The study drug will be administered with a subcutaneous injection of galcanezumab or placebo. The first dose (at month 1) will be a loading dose of two injections, or 240 mg in total. After that, at month 2 and month 3, each participant will get either a subcutaneous injection of galcanezumab 120 mg or placebo. The injections will be with a pre-loaded syringe containing either galcanezumab or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The following study procedures will be in place to ensure double-blind administration of study treatments. Access to the randomization code will be strictly controlled and this will reside with our pharmacist, who will not be blinded. All members of the clinical team and biostatistician will be blinded. Packaging and labeling of test and control treatments will be identical to maintain the blind. Each participant will be given an identical study packet, containing their assigned drug and study information. The study blind will be broken on completion of the clinical study and after the study database has been locked. Investigators will be made aware of their participants' treatment designations only after all the data has been collected and analyzed. During the study, the blind may be broken only in emergencies when knowledge of the participant's treatment group is necessary for further clinical management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galcanezumab (Experimental): The galcanezumab arm will self-administer a subcutaneous injection of galcanezumab. The first dose (at month 1) will be a loading dose of two injections, or 240 mg in total. After that, at month 2 and month 3, each participant will receive an injection of galcanezumab 120 mg. The injections will be with a pre-loaded syringe containing galcanezumab.
  Interventions: Drug: Galcanezumab Prefilled Syringe
- Placebo (Placebo Comparator): The placebo arm will self-administer a subcutaneous injection of placebo. The first dose (at month 1) will be a loading dose of two injections, or 240 mg in total. After that, at month 2 and month 3, each participant will receive an injection of placebo 120 mg. The injections will be with a pre-loaded syringe containing placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab Prefilled Syringe — Galcanezumab will be supplied in preloaded syringes, each with a dose of 120 mg. Participants will first receive the first month's supply (240 mg) at study visit 2, and then will receive a two month supply at study visit 3. So, at study visit 2 and 3, each participant will get two pre-filled syringes.
  Other Names: Emgality
  Arms: Galcanezumab
Drug: Placebo — Placebo will be supplied in preloaded syringes, each with a dose of 120 mg. Participants will first receive the first month's supply (240 mg) at study visit 2, and then will receive a two month supply at study visit 3. So, at study visit 2 and 3, each participant will get two pre-filled syringes.
  Arms: Placebo

SUMMARY:
Vestibular migraine (VM) has been recognized a distinct subtype of migraine that causes dizziness as the predominant symptom. Criteria for diagnosis have been adopted by the Barany Society. Previous epidemiological research from the investigators has shown that VM affects 2.7% of the adult population of the United States. Yet, despite its high prevalence, there is very little data upon which to guide treatment decisions. A Cochrane review in 2015 concluded that there were no placebo controlled trials in VM, and none have been done since then. The investigators recently developed and validated a patient reported outcome tool for VM called VM-PATHI (VM- Patient Assessment Tool and Handicap Inventory). Anecdotal evidence suggests that CGRP antagonists, such as Galcanezumab, may be effective in reducing or eliminating symptoms in VM. Therefore, the investigators propose a pilot study of changes in VM-PATHI scores, comparing active treatment (Galcanezumab) to placebo arms.

DETAILED DESCRIPTION:
Vestibular migraine (VM) is a distinct subtype of migraine that causes episodic vertigo/dizziness, sometimes with headache, and sometimes without. However, unlike traditional migraines, patients generally seek out care because of dizziness, and not because of headache. Therefore, these patients are cared for by a variety of providers who treat dizziness, including otolaryngologists and neurologists. Lifetime prevalence of VM in the general population is estimated to be 2.7%, and at least 10% of patients in a tertiary care vestibular clinic have VM. Furthermore, VM has been shown to decrease quality of life in multiple domains, including overall health, mental health, and emotional health. Since testing and imaging are usually normal, diagnosis can only be made on clinical grounds. Recently, consensus criteria for diagnosis was published by the Barany Society and the International Classification of Headache Disorders.

Galcanezumab is a calcitonin gene related peptide (CGRP) antagonist that has been approved by the FDA for treatment of episodic and chronic migraine. Its effects with regards to VM have not been formally studied. However, there is ample evidence to suggest that aberrant trigeminovascular inflammation may be integral to the pathophysiology of VM, similar to migraine in general.

This pilot study will be a single center, randomized double-blinded placebo-controlled trial comparing galcanezumab to placebo for treatment of VM. Screening data will be reviewed to determine subject eligibility. Participants who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. Participants in the galcanezumab arm will receive 240 mg via subcutaneous injection with a pre-loaded syringe at month 1, followed by 120 mg at month 2, and 120 mg at month 3. Those in the placebo arms will receive subcutaneous injections at the same time intervals of placebo. Randomization will occur through the hospital research pharmacy. Allocation concealment will be ensured; study participants will be given an envelope from a folder of sequentially ordered identical envelopes that will contain study instructions and the allocated drug. The master file linking study ID with allocation will be created by a third party and kept secret until after data analysis is complete. This will ensure that both providers and participants are adequately blinded. Blocking will be used in increments of 10 subjects to ensure equitable distribution of subjects into the two treatment arms. In addition, stratification by sex and definite versus probable vestibular migraine status will be used to ensure equal allocation. Total duration of subject participation will be five months. Total duration of the study is expected to be 2 years.

Data collection will be performed by the clinical research coordinator during each study visit. This data will be entered into the REDCap database by the research coordinator. VM- Patient Assessment Tool and Handicap Inventory (VM-PATHI), dizziness handicap inventory (DHI), General Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), Patient-Reported Outcomes Measurement Information System Short Form (PROMIS SF) v1.1- Global Health, and Headache Impact Test-6 (HIT-6) will be administered electronically via REDCap to the subject during the study visit.

There will be no stopping rules for this trial, given the short duration of the study. Each adverse effect and serious adverse effect will be reviewed by the data safety monitoring team, and subjects may be unblinded and/or the study will be stopped early for serious safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years of age at Study Visit 1.
2. Documentation of a vestibular migraine or probable vestibular migraine diagnosis according to the following criteria determined by the Barany Society:

   * Vestibular migraine

     * A: At least 5 episodes with vestibular symptoms of moderate or severe intensity, lasting 5 min to 72 hours
     * B: Current or previous history of migraine with or without aura according to the International Classification of Headache Disorders (ICHD)
     * C: One or more migraine features with at least 50% of the vestibular episodes:

       * Headache with at least two of the following characteristics: one sided location, pulsating quality, moderate or severe pain intensity, aggravation by routine physical activity
       * Photophobia and phonophobia
       * Visual aura
     * D: Not better accounted for by another vestibular or ICHD diagnosis
   * Probable vestibular migraine

     * At least 5 episodes with vestibular symptoms of moderate or severe intensity, lasting 5 min to 72 hours
     * Only one of the criteria B and C for vestibular migraine is fulfilled (migraine history or migraine features during the episode)
     * Not better accounted for by another vestibular or ICHD diagnosis
3. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
4. Baseline and Study Visit 2 VM-PATHI score > 25
5. Baseline (month 0 to 1) definite dizzy days > 4
6. Fluency in English
7. 80% adherence or better to daily text message during baseline phase
8. Written informed consent
9. Access to email, and cell phone

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to use approved form of birth control during participation in the study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Allergy to galcanezumab
4. Prior treatment with galcanezumab
5. History of ear surgery (other than ear tubes)
6. Other vestibular diagnosis (excluding treated Benign Paroxysmal Positional Vertigo- BPPV). This includes Meniere's disease, superior canal dehiscence syndrome, vestibular neuritis, persistent postural perceptual dizziness, unilateral or bilateral vestibular loss, cerebellar or brainstem disease, multiple sclerosis, or Mal de Debarquement.
7. Failure of treatment with > 4 prophylactic migraine medications
8. Prior or current treatment with a CGRP medication
9. Pregnant/breastfeeding if female
10. History of serious medical or psychiatric disease, at the discretion of the treating physician (including significant coronary artery disease, peripheral vascular disease, cerebrovascular disease, kidney disease, liver disease, Raynaud's disease, uncontrolled psychiatric disease or past psychiatric hospitalization)
11. History of mania, psychosis, or suicidal ideations
12. Ok if on up to 2 migraine prophylactic medications (prescribed for that purpose), dose must be stable for 2 months prior to study start.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Sharon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Mount Zion, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Ombergen A, Van Rompaey V, Van de Heyning P, Wuyts F. Vestibular migraine in an otolaryngology clinic: prevalence, associated symptoms, and prophylactic medication effectiveness. Otol Neurotol. 2015 Jan;36(1):133-8. doi: 10.1097/MAO.0000000000000596. PMID 25251304
- [Background] Formeister EJ, Rizk HG, Kohn MA, Sharon JD. The Epidemiology of Vestibular Migraine: A Population-based Survey Study. Otol Neurotol. 2018 Sep;39(8):1037-1044. doi: 10.1097/MAO.0000000000001900. PMID 30020261
- [Background] Lempert T, Olesen J, Furman J, Waterston J, Seemungal B, Carey J, Bisdorff A, Versino M, Evers S, Newman-Toker D. Vestibular migraine: diagnostic criteria. J Vestib Res. 2012;22(4):167-72. doi: 10.3233/VES-2012-0453. PMID 23142830
- [Background] Furman JM, Marcus DA, Balaban CD. Vestibular migraine: clinical aspects and pathophysiology. Lancet Neurol. 2013 Jul;12(7):706-15. doi: 10.1016/S1474-4422(13)70107-8. PMID 23769597
- [Background] Vass Z, Dai CF, Steyger PS, Jancso G, Trune DR, Nuttall AL. Co-localization of the vanilloid capsaicin receptor and substance P in sensory nerve fibers innervating cochlear and vertebro-basilar arteries. Neuroscience. 2004;124(4):919-27. doi: 10.1016/j.neuroscience.2003.12.030. PMID 15026132
- [Background] Salviz M, Yuce T, Acar H, Karatas A, Acikalin RM. Propranolol and venlafaxine for vestibular migraine prophylaxis: A randomized controlled trial. Laryngoscope. 2016 Jan;126(1):169-74. doi: 10.1002/lary.25445. Epub 2015 Jul 30. PMID 26228645
- [Background] Reploeg MD, Goebel JA. Migraine-associated dizziness: patient characteristics and management options. Otol Neurotol. 2002 May;23(3):364-71. doi: 10.1097/00129492-200205000-00024. PMID 11981397
- [Background] Mikulec AA, Faraji F, Kinsella LJ. Evaluation of the efficacy of caffeine cessation, nortriptyline, and topiramate therapy in vestibular migraine and complex dizziness of unknown etiology. Am J Otolaryngol. 2012 Jan-Feb;33(1):121-7. doi: 10.1016/j.amjoto.2011.04.010. Epub 2011 Jun 24. PMID 21704423
- [Background] Lepcha A, Amalanathan S, Augustine AM, Tyagi AK, Balraj A. Flunarizine in the prophylaxis of migrainous vertigo: a randomized controlled trial. Eur Arch Otorhinolaryngol. 2014 Nov;271(11):2931-6. doi: 10.1007/s00405-013-2786-4. Epub 2013 Oct 29. PMID 24166742
- [Background] Maldonado Fernandez M, Birdi JS, Irving GJ, Murdin L, Kivekas I, Strupp M. Pharmacological agents for the prevention of vestibular migraine. Cochrane Database Syst Rev. 2015 Jun 21;2015(6):CD010600. doi: 10.1002/14651858.CD010600.pub2. PMID 26093662
- [Result] Sharon JD, Krauter R, Chae R, Gardi A, Hum M, Allen I, Levin M. A placebo controlled, randomized clinical trial of galcanezumab for vestibular migraine: The INVESTMENT study. Headache. 2024 Nov-Dec;64(10):1264-1272. doi: 10.1111/head.14835. Epub 2024 Sep 30. PMID 39344988

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Galcanezumab | Placebo
Started | 18 | 22
Completed | 17 | 21
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — study unexpectedly stopped early due to supply issues with drug/placebo | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galcanezumab | Placebo | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.0) | 47.3 (14.5) | 50.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 4 | 6 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 16 | 30
  Asian | 1 | 2 | 3
  Black | 1 | 0 | 1
  Other | 2 | 4 | 6
History of migraine [Count of Participants; unit: Participants] | 17 | 20 | 37
Family history of migraine [Count of Participants; unit: Participants] | 11 | 13 | 24
Count of triggers [Mean (Standard Deviation); unit: Count of triggers] | 9.4 (7.8) | 8.9 (7.6) | 9.1 (3.0)
Count of associated symptoms [Mean (Standard Deviation); unit: count of associated symptoms] | 4.2 (1.7) | 4.6 (1.3) | 4.4 (1.5)
SV2 VM-PATHI score [Mean (Standard Deviation); unit: mean score] — This the VM-PATHI (Vestibular Migraine Patient Assessment Tool and Handicap Inventory) score for Study Visit 2 (SV2). VM-PATHI is a scale measure symptom severity in vestibular migraine. Scores range from 0 (no symptoms) to 100 (worst score possible indicating severe symptoms). The numbers represent the total score for the VM-PATHI.
  mean score | 47.3 (12) | 45.7 (9.9) | 46.4 (10.8)
SV2 DHI score [Mean (Standard Deviation); unit: mean score] — This is the Dizziness Handicap Inventory (DHI) score for Study Visit 2 (SV2). DHI scores represent how severely dizziness is affecting someone. Scores range from 0 (no effect), to 100 (the most severe effect possible). The number is the total score on the DHI.
  mean score | 61.4 (14.9) | 56.7 (19.1) | 58.8 (17.3)
DDD baseline [Mean (Standard Deviation); unit: days] — DDD is a Definitive Dizzy Day. Each day during the baseline period, participants were texted, and they had to response to a question inquiring about their level of dizziness during the prior 24 hours. Answer choices included none (0), mild (1), moderate (2), and severe (3). A score of 2 or 3 was counted as a DDD. Therefore, this shows the count of DDDs during the baseline month.
  days | 17.9 (7.9) | 18 (7.6) | 18 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in VM-PATHI (Vestibular Migraine-Patient Assessment Tool and Handicap Inventory) Score From Baseline to Month 4
Description: This is a recently developed and validated outcome measure for vestibular migraine from the investigators. It has been shown to be highly reliable and valid, and responsive to treatment changes. At this point, it is the only disease specific outcome measure for vestibular migraine. Scores are between 0 and 100, with 100 indicating higher levels of disease related suffering.
Time Frame: Change between baseline (month 1) and after treatment (month 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galcanezumab | Placebo
Number analyzed (Participants) | 17 | 21
score on a scale | -14.8 (16.1) | -5.1 (17.3)

2. Secondary Outcome: Change in Number of Definitive Dizzy Days for Participants Measured Daily From Baseline to Month 4 Via Text Message
Description: Participants will receive a daily text message to rate their dizziness from 0 (no dizziness), 1 (mild dizziness), 2 (moderate dizziness), and 3 (severe dizziness). A score of 2 or higher will count as a definitive dizzy day.
Time Frame: Change between baseline (month 0) and after treatment (month 4)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Galcanezumab | Placebo
Number analyzed (Participants) | 17 | 21
days | -11.3 (7.2) | -5.6 (7.9)

3. Secondary Outcome: Change in Response Rates as Defined by Percentage Reduction in Definitive Dizzy Days Via Text Message From Baseline to Month 4
Description: Response rates will be measured by the percentage of participants in each arm experiencing a 100%, 75%, 50%, 25%, 0% reduction in definitive dizzy days.
Time Frame: Change between baseline (month 0) to after treatment (month 4)
Measure: Number; unit: percentage of subjects
Arm/Group | Galcanezumab | Placebo
Number analyzed (Participants) | 17 | 21
percentage of subjects
  100% reduction | 18 | 10
  75% reduction | 53 | 38
  50% reduction | 77 | 48
  25% reduction | 82 | 57

4. Secondary Outcome: Change in Dizziness Handicap Inventory Score From Baseline to Month 4
Description: This is the most widely used measure of dizziness severity, and consists of 25 questions. Questions ask about problems related to dizziness, and are scored as no (0 points), sometimes (2 points), or always (4 points). Total score is between 0 and 100, with higher scores indicating more disability.
Time Frame: Change between baseline (month 0) to after treatment (month 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Galcanezumab | Placebo
Number analyzed (Participants) | 17 | 21
score on a scale | -22 (19.3) | -8.3 (15)

5. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System Short Form (PROMIS SF) v1.2- Global Health Scores
Description: There are 10 questions on this quality of life measure, each with a score of 1-5. Higher scores correspond to a greater extent of the concept measured (e.g., more fatigue). Two summed scores are generated, one for global mental health (question #3, 6, 7, 8) and one for global physical health (question #2, 4, 5, 10). The remaining 2 questions are analyzed separately.
  Summed scores for physical health and mental health are converted into T-score values using the "HealthMeasures Scoring Service" available online.
  The average score for the US population is 50, with a standard deviation of 10. Higher scores indicate better physical and mental health.
Time Frame: Change between baseline (month 1) to after treatment (month 4)
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Galcanezumab | Placebo
Number analyzed (Participants) | 17 | 21
t score
  physical subscale | 5.3 (7) | 1.9 (6.4)
  mental subscale | 4.8 (5.3) | 3.2 (8.3)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Galcanezumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 4/18 | 8/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galcanezumab (N=18) | Placebo (N=22)
injection site reaction (Skin and subcutaneous tissue disorders) | 2 | 0
worsening of vestibular migraines (Nervous system disorders) | 2 | 0
injection site soreness (Skin and subcutaneous tissue disorders) | 0 | 1
injection site bruising (Skin and subcutaneous tissue disorders) | 0 | 1
subjective weight gain (Metabolism and nutrition disorders) | 0 | 1
low blood pressure (Vascular disorders) | 0 | 1
increased headaches (Nervous system disorders) | 0 | 1
hair loss (Skin and subcutaneous tissue disorders) | 0 | 1
palpitations (Cardiac disorders) | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04417361/Prot_SAP_001.pdf